CLINICAL TRIAL: NCT04107844
Title: Safe Return to Play After Concussion, Increased Knowledge of a Potential Physiological Deficit After Cessation of Symptoms
Brief Title: Safe Return to Play After Concussion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College of Northern Denmark (Other)
Responsible Party: Principal Investigator, Signe Refsgaard Bech, Associate Professor, Ph.d., University College of Northern Denmark
Other Study IDs: Concussiondualtask
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Concussion, Brain; Sports Injury
Keywords: return to play; pain catastrophizing; athletes
MeSH Terms: conditions — Brain Concussion; Athletic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes without concussion: We follow the athletes in terms of injuries and make a baseline test each season.
  Interventions: Diagnostic Test: Novel facilitating agility dual-task test combined with already known tests
- Athletes suffering a concussion: We follow the athletes in terms of injuries and make a baseline test each season and when they suffer a concussion, then we follow them with the same test as at baseline every 14th day for 3 months, after that they will get enrolled in another study.
  Interventions: Diagnostic Test: Novel facilitating agility dual-task test combined with already known tests

INTERVENTIONS:
Diagnostic Test: Novel facilitating agility dual-task test combined with already known tests — We will investigate if a combination of a novel Dual-task test combined with already known tests can identify more athletes, not ready to return to play, although symptoms of concussion have stopped.

SUMMARY:
This study will evaluate a combination of a novel Dual-task regime together with other already known tests in terms of defining when an athlete is ready to return to play after a concussion.

DETAILED DESCRIPTION:
In this prospective study, we will evaluate a combination of a novel facilitating agility Dual-task regime together with sport concussion assessment tool -5 (SCAT5), Vestibular/Ocular-Motor Screening for Concussion, Agility T-test, Joint repositions error test and Pain Catastrophizing Scale (PCS) in terms of defining when an athlete is ready to return to play after a concussion. We will investigate if a novel facilitating agility Dual-task test together with already widely used tests, can identify more athletes that after a concussion still isn't ready to return to play, due to a physiological deficit. We will test as many athletes as possible each season and when an athlete suffer a concussion, we will follow them to see when they reach their baseline level. As previous studies show a over representation of new injuries in athletes returning to play after a concussion, we will also register injuries from all included subjects in terms of injuries each year, to evaluate if athletes following our recommendations have a lower injury rate after returning to play after a concussion. We also hope to be able to get more knowledge about how pain catastrophizing is related to duration of concussions symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Athletes participating in sports at least 1xweek

Exclusion Criteria:

* injury that limits the participants ability to conduct the tests If the participant don't speak and understand Danish or English Other diseases or conditions that could interfere with one or more of the tests.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Athletes participating in risk sports in terms of concussion.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Duration from concussion to physiological rehabilitated with a combination of new and already known test evaluate when the athlete is ready to return to play. | as it is a prospective study and we don't know when and how many athletes will get a concussion, then the timeframe is unknown, but we expect to collect data in at least 4 years.
  We will by using a combination of new and known tests follow athletes with concussion and their symptoms, and try to get a knowledge about easy accessable test can give coaches a more objective measure for when an athlete is ready to return to play.

SECONDARY OUTCOMES:
How pain catastrophizing influence recovery after a concussion | at least 4 years
  Be measuring pain catastrophizing at baseline and after concussion, we will evaluate if pain catastrophizing correlates with recovery time.

CONTACTS AND LOCATIONS:
Overall Officials: Signe R Bech, Phd, Principal Investigator — University College of Northern Denamrk
Locations (1):
- Signe Refsgaard Bech, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Maybe we will share data on the concussed athletes.